CLINICAL TRIAL: NCT00195364
Title: Long-Term Safety Study of Etanercept in Patients With Rheumatoid Arthritis Who Completed Trial 0881A1-301-EU in Spain
Brief Title: Study Evaluating Etanercept in Patients With Rheumatoid Arthritis Who Completed Trial 0881A1-301-EU in Spain
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0881A1-301, 101492
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Rheumatoid Arthritis; Inflammation
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to evaluate long-term safety of etanercept in patients with rheumatoid arthritis who successfully have completed open-label safety study 0881A1-301-EU

ELIGIBILITY:
Inclusion Criteria:

* To have completed 0881A1-301-EU study in Spain
* Clinical diagnosis by ACR revised criteria of rheumatoid arthritis.

Exclusion Criteria:

* Hypersensibility to etanercept or any of its components
* Significant concurrent medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who completed trial 0881A1-301-EU in Spain who fulfill inclusion/exclusion criteria, treated in rheumatology units
Sampling Method: Probability Sample
Enrollment: 93
Dates: Start 2003-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Madrid, Madrid, Spain